CLINICAL TRIAL: NCT04805203
Title: Analysis of the Immune Parameters Involved in the Onset and Fate of SARS-CoV-2 Infection in Patients With Multiple Myeloma (COVIMMUNOMM) COVID-19 and Multiple Myeloma
Brief Title: Analysis of the Immune Parameters of COVID-19 Infection in Patients With Multiple Myeloma
Acronym: Covimmunomm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment delay due to difficulties to involve patient at Covid diagnosis in hematology departments Abandoned study
Sponsor: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IFM 2020-08
Record Dates: First submitted 2020-12-15; First posted 2021-03-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma; Covid19
Keywords: Multiple Myeloma; Covid19
MeSH Terms: conditions — Multiple Myeloma; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood samples (Other): 4 blood samples per patient maximum (at diagnosis of covid19, during intensive care if applicable, at revecory of covid 19 and 6 months after recovery.
  Interventions: Other: blood sample analyses

INTERVENTIONS:
Other: blood sample analyses — maximum 4 blood samples analyses per patient. At diagnosis of covid 19, in intensif care (if applicable), at covid19 recovery and 6 months after recovery

SUMMARY:
Among all MM patients included in the cohort at the time of diagnosis of SARS-CoV-2 infection, blood samples will be collected at inclusion, at time of the infection acute phase in the most severe cases (when admitted in intensive care units), and at recovery. The following immune function tests will be evaluated, gammaglobulin measurements, lymphocytes counts, B, T, and NK cells analyses by cytometry, including exhaustion analyses. In addition, T cell repertoire sequencing looking for SARS-CoV-2- specific T cells, and serologies, will be evaluated at recovery and 6 months after MM treatment re-initiation.

DETAILED DESCRIPTION:
MM is a hematological malignancy, supposed mainly not curable, except for some exceptional patients, despite the availability of numerous new drugs. The patients are highly susceptible to infections, both bacterial and viral, due to a defect immune status, both at the antibody level (hypogammaglobulinemia) and the cellular level. This immunosuppression is further worsened by the treatments, and especially high dose glucocorticoids used at each phase of the disease. Consequently, MM patients are highly susceptible to contract COVID19, and to develop a severe form. This has been confirmed in a first study in Spring, showing a mortality rate of 37%. Among all MM patients included in the cohort at the time of diagnosis of SARS-CoV-2 infection, blood samples will be collected at inclusion, at time of the infection acute phase in the most severe cases (when admitted in intensive care units), and at recovery. The following immune function tests will be evaluated, gammaglobulin measurements, lymphocytes counts, B, T, and NK cells analyses by cytometry, including exhaustion analyses. In addition, T cell repertoire sequencing looking for SARS-CoV-2- specific T cells, and serologies, will be evaluated at recovery and 6 months after MM treatment re-initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a multiple myeloma and a documented COVID19 (by RT-PCR, thoracic TDM, and/or antigenix test).
* Patients having received the information to participate in the research and having expressed their non-opposition
* Patients with social security insurance or equivalent

Exclusion Criteria:

* Patients without multiple myeloma
* Patients without COVID19
* Patients under juridical protection guardianship, or tutelage measure

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Characterize the immune laboratory parameters of Multiple Myeloma patients at the start of infection with COVID-19 | up to one month following COVID-19 diagnosis
  gammaglobulin measurements in g/L
Characterize the immune laboratory parameters of Multiple Myeloma patients at the cure of COVID-19 | one month following COVID-19 diagnosis
  gammaglobulin measurements in g/L
Characterize the immune laboratory parameters of Multiple Myeloma patients at the start of infection with COVID-19 | up to one month following COVID-19 diagnosis
  lymphocytes counts in g/l
Characterize the immune laboratory parameters of Multiple Myeloma patients at the cure of COVID-19 | one month following COVID-19 diagnosis
  lymphocytes counts in g/l
Characterize the immune laboratory parameters of Multiple Myeloma patients at the start of infection with COVID-19 | up to one month following COVID-19 diagnosis
  number of cells B, T, and NK actived and inhibited
Characterize the immune laboratory parameters of Multiple Myeloma patientsat the cure of COVID-19 | one month following COVID-19 diagnosis
  number of cells B, T, and NK actived and inhibited
Correlation of patient immune function with death or development of protective immunity | up to 6 months following COVID-19 diagnosis
  number of death

SECONDARY OUTCOMES:
Number of patient with protective immune response | before the reintroduction of MM treatments, and 6 months later to evaluate if those treatments
  T cell repertoire sequencing looking for SARS-CoV-2- specific T cells, and serologies

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Avet Loiseau, PU-PH, Principal Investigator — Intergroupe Francophone du Myelome
Locations (53):
- France (53):
  - CHU Amiens SUD, Amiens
  - CHRU Hôpital du Bocage, Angers
  - Ch Annecy Genevois, Annecy
  - CH Victor Dupouy, Argenteuil
  - CH d'ARRAS, Arras
  - CH Auch, Auch
  - Centre Hospitalier H.Duffaut, Avignon
  - CHRU Besançon, Besançon
  - Centre Hospitalier Simone Veil de Blois, Blois
  - CHU Bordeaux-hopital haut leveque, Bordeaux
  - Centre hospitalier Pierre Oudot, Bourgoin
  - Hôpital A.Morvan, Brest
  - CHU de Caen, Caen
  - CH de Cannes, Cannes
  - Clinique du Parc, Castelnau-le-Lez
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier Métropole de Savoie, Chambéry
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CH de Dax côte d'Argent, Dax
  - CHU François Mitterand, Dijon
  - CHU grenoble, Grenoble
  - Institut Daniel Hollard - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CH de Lens, Lens
  - Hopital Claude Huriez-CHRU LILLE, Lille
  - CHU Limoges, Limoges
  - Centre Hospitalier Lyon sud, Lyon
  - GHT des Landes, Mont-de-Marsan
  - CHU saint Eloi, Montpellier
  - Hôpital E. MULLER, Mulhouse
  - Hôpitaux de Brabois - CHRU de Nancy, Nancy
  - CHRU Nantes, Nantes
  - Hopital Archet 1, Nice
  - Hopital Cochin, Paris
  - Hopital Saint Antoine, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - CHU de Reims, Reims
  - Chu Pontchaillou, Rennes
  - CH Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest
  - Centre Hospitalier, Saint-Quentin
  - ICANS, Strasbourg
  - CH Tarbes, Tarbes
  - CHU Toulouse, Toulouse
  - CHRU Bretonneau, Tours
  - CH de valenciennes, Valenciennes
  - CH Bretagne Atlantique Vannes et Auray-P.Chubert, Vannes
  - CHV André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: No